CLINICAL TRIAL: NCT05721066
Title: Hemostatic Profile of Post COVID-19/Long COVID-19 Patients
Acronym: LCV
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Dr, IRCCS Policlinico S. Donato
Other Study IDs: LONG-COVID-VET
Record Dates: First submitted 2023-02-08; First posted 2023-02-09 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Post-acute COVID-19 Syndrome
Keywords: COVID-19; Post-acute COVID-19 Syndrome; Coagulopathy; Fibrinolysis; Thrombosis
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Hemostatic Disorders; Thrombosis | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POST-COVID: Patients hospitalized due to acute COVID-19 pneumonia and discharged home. No residual symptoms after recovery. Contacted by phone and invited to an in-person interview about their health conditions and a blood withdrawal for the assessment of the coagulation profile (both in standard laboratory and point-of-care device ClotPro).
  Interventions: Diagnostic Test: ClotPro assessment; Diagnostic Test: Laboratory analysis; Other: Interview
- LONG-COVID: Patients hospitalized due to acute COVID-19 pneumonia and discharged home. Presence of residual symptoms after recovery or new symptoms appeared after discharge not otherwise explained.
  Contacted by phone and invited to an in-person interview about their health conditions and a blood withdrawal for the assessment of the coagulation profile (both in standard laboratory and point-of-care device ClotPro).
  Interventions: Diagnostic Test: ClotPro assessment; Diagnostic Test: Laboratory analysis; Other: Interview

INTERVENTIONS:
Diagnostic Test: ClotPro assessment — Point-of-care viscoelastic assessment of the coagulation profile (extrinsic pathway, intrinsic pathway, fibrinogen contribution, tPA stimulated fibrinolysis)
Diagnostic Test: Laboratory analysis — Blood count and standard coagulation tests (INR, aPTT, fibrinogen, D-dimers, antithrombin)
Other: Interview — Questionnaire from ISS (Istituto Superiore Sanità, the National Health Institute) about the health conditions before the acute COVID-19 infection, the disease (and the hospitalization) details and the eventual health disturbances experienced after the recovery from COVID-19 infection.

SUMMARY:
The present study aims at assessing long-term hemostatic profile of patients recovered from COVID-19 acute infection that remain asymptomatic (POST-COVID) versus patients with residual symptoms (LONG-COVID) through the employment of a commercially available new generation point-of-care viscoelastic device. The primary endpoint is based upon the hypothesis that patients with residual symptoms maintain an abnormal coagulation profile even after recovery from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* recovery from acute COVID-19 infection;
* COVID-19 pneumonia that required hospitalization in our Institution;
* discharge from the hospital minimum 3 months before the day of the visit;
* written consent to participate to the study.

Exclusion Criteria:

* none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The list of the patients hospitalized in our Institution due to COVID-19 pneumonia (positive COVID-19 test and radiological pneumonia diagnosis) was retrieved. The patients were recruited through a phone contact, those who were reachable and agreed to participate received an appointment for the in-person study-related procedures at our Hospital. The eligible patient population was represented by subjects hospitalized at out Institution for COVID-19 infection between January 1, 2021, and July 31, 2022. The planned patient population was 100 patients. The final patient population comprised 102 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
ClotPro EXTEST | Day of the visit
  Extrinsic pathway of the coagulation as measured by the ClotPro (coagulation time CT, seconds; maximum clot firmness, MCF, millimeters)
ClotPro INTEST | Day of the visit
  Intrinsic pathway of the coagulation as measured by the ClotPro (coagulation time CT, seconds; maximum clot firmness, MCF, millimeters)
ClotPro FIBTEST | Day of the visit
  Fibrinogen contribution to the overall clot strength as measured by the ClotPro (maximum clot firmness, MCF, millimeters)
ClotPro TPATEST | Day of the visit
  Resistance to the fibrinolysis induced by the tPA (tissue plasminogen) as measured by the ClotPro (lysis time, LT, seconds; maximum lysis, ML, %).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The original dataset supporting the findings of this study will be deposited in the public repository Zenodo after the publication of the paper and accessible upon a reasonable request to the Principal Investigator.